CLINICAL TRIAL: NCT00667225
Title: Efficacy of Cantharidin in Molluscum Contagiosum: A Randomized, Blinded, Placebo-Controlled Prospective Study
Brief Title: Efficacy of Cantharidin in Molluscum Contagiosum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); Doris Duke Charitable Foundation (Other)
Responsible Party: Jacquelyn Coloe, Doris Duke Clinical Research Fellow, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB 07-1330; RR000046 (Other Grant/Funding Number: National Center for Research Resources (NCRR))
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2011-06-01 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Molluscum Contagiosum, Skin Disease
MeSH Terms: conditions — Molluscum Contagiosum; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Placebo Comparator): Subjects in this group will have topical application of cantharidin's vehicle at each visit.
  Interventions: Drug: cantharidin's vehicle
- II (Experimental): Subjects in this group will have topical application of cantharidin at each visit.
  Interventions: Drug: Cantharidin 0.7%

INTERVENTIONS:
Drug: cantharidin's vehicle — Cantharidin's vehicle is composed of: Hydroxypropylcellulose, Acetone, and Collodion Flexible. The vehicle will be topically applied to molluscum lesions at each visit. Only two lesions will be treated at the first visit, and up to 20 lesions can be treated at subsequent visits.
  Arms: I
Drug: Cantharidin 0.7% — Subjects in this arm will receive cantharidin at all visits. At the first visit, up to 2 lesions can have application with cantharidin. All other visits will have up to 20 lesions with application of the cantharidin. During every visit, lesions will be counted and subjects will be assessed for any adverse events.
  Arms: II

SUMMARY:
The University of North Carolina Department of Dermatology is conducting a clinical trial to evaluate a drug called cantharidin in the treatment of molluscum contagiosum. Molluscum is a common dermatologic disorder caused by a poxvirus. Molluscum typically presents with many flesh-colored bumps on the skin. It goes away on its own, though can last several months to several years. Cantharidin is a topical medicine which is applied at the clinic visit. It is well tolerated by the majority of children.

ELIGIBILITY:
Inclusion Criteria:

* Anyone aged 5-10 years with the clinical diagnosis of molluscum contagiosum.

Exclusion Criteria:

* Anyone with immunosuppression including HIV or previous organ transplantation.
* Anyone taking immunosuppressive medications.
* Anyone who has previously received treatment with cantharidin.
* Any female who has had her first menstrual period.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2008-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacquelyn R Dosal, MD, Principal Investigator — UNC
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the UNC Dermatology clinics, through practitioners in the surrounding community, and through mass email to the University system (University of Chapel Hill).
Pre-assignment Details: Participants were excluded if they did not meet inclusion criteria, if they did not have a true diagnosis of molluscum contagiosum, if they were immunosuppressed, or if they had previously been treated with cantharidin.
Groups:
- Vehicle: Subjects in this group will have topical application of cantharidin's vehicle at each visit. Vehicle will be applied every two weeks for a total of 5 visits (4 applications, one follow up visit, for a total of 8 weeks). The solution is applied topically with the stick end of a cotton tipped applicator to the lesion with care to avoid normal skin. Up to 2 lesions were treated on the first visit, and up to 20 lesions were treated on subsequent visits. Parents were instructed to wash the area 4 hours after application.
- Cantharidin: Subjects in this group will have topical application of cantharidin at each visit. Cantharidin will be applied every two weeks for a total of 5 visits (4 applications, one follow up visit, for a total of 8 weeks). The solution is applied topically with the stick end of a cotton tipped applicator to the lesion with care to avoid normal skin. Up to 2 lesions were treated on the first visit, and up to 20 lesions were treated on subsequent visits. Parents were instructed to wash the area 4 hours after application.
Period: Overall Study
Arm/Group | Vehicle | Cantharidin
Started | 16 | 13
Completed | 15 | 12
Not Completed | 1 | 1
Not completed — Subject had no more lesions to treat. | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle | Cantharidin | Total
Number analyzed (Participants) | 16 | 13 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 13 | 29
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 7.3 (1.7) | 6.7 (1.8) | 7 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 16 | 13 | 29

OUTCOME MEASURES:

1. Primary Outcome: Patients Experiencing Complete Clearance of All Molluscum Lesions.
Time Frame: Baseline compared to 8 weeks (5 visits)
Population: We used a power calculation to estimate the number of patients needed to detect a clinically significant result.
Measure: Number; unit: Participants
Units Other Than Participants: Participants
Arm/Group | Vehicle | Cantharidin
Number analyzed (Participants) | 16 | 13
Participants | 1 | 3

2. Secondary Outcome: Mean Change in Each Group Measured by Lesion Count.
Description: Average change in number of lesions from baseline to 8 weeks
Time Frame: Baseline compared to 8 weeks (5 visits)
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Vehicle | Cantharidin
Number analyzed (Participants) | 16 | 13
lesions | 26.26 (27.55) | 35.61 (48.15)

ADVERSE EVENTS:
Arm/Group | Vehicle | Cantharidin
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/13
Other Adverse Events (participants affected / at risk) | 1/16 | 3/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=16) | Cantharidin (N=13)
Pain after application of cantharidin or vehicle (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) — Self-reported pain after application. One patient in the cantharidin group reported pain with removal (with soap and water) of the medication.

LIMITATIONS AND CAVEATS:
Small sample size and random disproportionate assignment to the vehicle group. Other limitations include short duration of follow up and interval between treatments. Finally, matching subjects in each group with comparable lesion counts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No